CLINICAL TRIAL: NCT05970120
Title: Clinical Evaluation of Intracardiac Ultrasound With the NUVISION NAV Ultrasound Catheter
Brief Title: A Study of Intracardiac Ultrasound With the NUVISION NAV Ultrasound Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202104; BWI202104 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Scar-related Atrial Tachycardia; Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Ventricular Tachycardia; Premature Ventricular Complex
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NUVISION NAV Ultrasound Catheter (Experimental): Participants with five different subgroups (scar-related atrial tachycardia, persistent atrial fibrillation [PsAF], paroxysmal atrial fibrillation [PVF], ventricular tachycardia [VT], and premature ventricular complex [PVC]) will be treated using NUVISION NAV ultrasound catheter per investigator's standard of care and followed until 7 days post-procedure.
  Interventions: Device: NUVISION NAV Ultrasound Catheter

INTERVENTIONS:
Device: NUVISION NAV Ultrasound Catheter — Participants will be scheduled to have a clinically-indicated ablation procedure using NUVISION NAV ultrasound catheter for management of atrial procedure.

SUMMARY:
The purpose of this study is to assess the performance and safety of using the investigational catheter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with and candidate for clinically-indicated cardiac ablation procedure for the management of ventricular tachycardia, premature ventricular complex, scar-related atrial tachycardia or atrial fibrillation (participants having undergone a previous ablation procedure may be included)
* Signed participants Informed Consent Form (ICF)
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Structural heart defect which can only be repaired by cardiac surgery
* Pericarditis within 6 months
* Left ventricular ejection fraction (LVEF) less than or equal to (<=) 25 percent (%) for ventricular tachycardia (VT) participants
* LVEF <= 40% for participants with atrial arrhythmia
* History of chronic gastro-intestinal medical problems involving the esophagus, stomach and/or untreated acid reflux
* History of abnormal bleeding and/or clotting disorder
* Clinically significant infection or sepsis
* History of stroke or transient ischemic attack (TIA) within the past 6 months of enrollment
* Uncontrolled heart failure or New York Heart Association (NYHA) function class IV
* Implanted with a pacemaker or intracardiac cardiac defibrillator within the past 6 weeks (42 days)
* Implanted with a mechanical valve
* Diagnosed atrial or ventricular myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation
* Any of the following within 6 months of enrollment: major surgery except for the index procedure, myocardial infarction, unstable angina, percutaneous coronary intervention
* Participants with any other significant uncontrolled or unstable medical condition (such as uncontrolled bradyarrhythmia's, ventricular arrhythmias, hyperthyroidism, or significant coagulation disorder)
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of childbearing age and plan on becoming pregnant during the course of the clinical investigation
* Categorized as vulnerable population and requires special treatment with respect to safeguards of well-being
* Concurrent enrollment in an investigational study evaluating another device or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (3):
- KBC Split, Split, Croatia
- Yitzhak Shamir Medical Center, Ẕerifin, Israel
- Centro Cardiologico Monzino, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Perk G, Lang RM, Garcia-Fernandez MA, Lodato J, Sugeng L, Lopez J, Knight BP, Messika-Zeitoun D, Shah S, Slater J, Brochet E, Varkey M, Hijazi Z, Marino N, Ruiz C, Kronzon I. Use of real time three-dimensional transesophageal echocardiography in intracardiac catheter based interventions. J Am Soc Echocardiogr. 2009 Aug;22(8):865-82. doi: 10.1016/j.echo.2009.04.031. PMID 19647156
- [Background] Faletra FF, Pedrazzini G, Pasotti E, Muzzarelli S, Dequarti MC, Murzilli R, Schlossbauer SA, Slater IP, Moccetti T. 3D TEE during catheter-based interventions. JACC Cardiovasc Imaging. 2014 Mar;7(3):292-308. doi: 10.1016/j.jcmg.2013.10.012. PMID 24651102
- [Background] Anter E, Silverstein J, Tschabrunn CM, Shvilkin A, Haffajee CI, Zimetbaum PJ, Buxton AE, Josephson ME, Gelfand E, Manning WJ. Comparison of intracardiac echocardiography and transesophageal echocardiography for imaging of the right and left atrial appendages. Heart Rhythm. 2014 Nov;11(11):1890-7. doi: 10.1016/j.hrthm.2014.07.015. Epub 2014 Jul 14. PMID 25034183
- [Background] Rigatelli G, Dell'Avvocata F, Giordan M, Viceconte N, Osanna RA, Braggion G, Aggio S, Cardaioli P, Chen JP. Usefulness of intracardiac echocardiography with a mechanical probe for catheter-based interventions: a 10-year prospective registry. J Clin Ultrasound. 2014 Nov-Dec;42(9):534-43. doi: 10.1002/jcu.22177. Epub 2014 Jun 4. PMID 24898198
- [Background] Medford BA, Taggart NW, Cabalka AK, Cetta F, Reeder GS, Hagler DJ, Johnson JN. Intracardiac echocardiography during atrial septal defect and patent foramen ovale device closure in pediatric and adolescent patients. J Am Soc Echocardiogr. 2014 Sep;27(9):984-90. doi: 10.1016/j.echo.2014.05.017. Epub 2014 Jul 4. PMID 24998516
- [Background] Kabra R, Singh J. Recent trends in imaging for atrial fibrillation ablation. Indian Pacing Electrophysiol J. 2010 May 5;10(5):215-27. PMID 20473373
- [Background] Lee W, Griffin W, Wildes D, Buckley D, Topka T, Chodakauskas T, Langer M, Calisti S, Bergstol S, Malacrida JP, Lanteri F, Maffre J, McDaniel B, Shivkumar K, Cummings J, Callans D, Silvestry F, Packer D. A 10-Fr ultrasound catheter with integrated micromotor for 4-D intracardiac echocardiography. IEEE Trans Ultrason Ferroelectr Freq Control. 2011 Jul;58(7):1478-91. doi: 10.1109/TUFFC.2011.1967. PMID 21768032
- [Background] Silvestry FE, Kadakia MB, Willhide J, Herrmann HC. Initial experience with a novel real-time three-dimensional intracardiac ultrasound system to guide percutaneous cardiac structural interventions: a phase 1 feasibility study of volume intracardiac echocardiography in the assessment of patients with structural heart disease undergoing percutaneous transcatheter therapy. J Am Soc Echocardiogr. 2014 Sep;27(9):978-83. doi: 10.1016/j.echo.2014.04.022. Epub 2014 Jun 11. PMID 24930123
- [Background] Alkhouli M, Chaker Z, Alqahtani F, Raslan S, Raybuck B. Outcomes of Routine Intracardiac Echocardiography to Guide Left Atrial Appendage Occlusion. JACC Clin Electrophysiol. 2020 Apr;6(4):393-400. doi: 10.1016/j.jacep.2019.11.014. Epub 2020 Jan 29. PMID 32327072
- [Background] Flautt T, Da-Wariboko A, Lador A, Patel A, Guevara M, Valderrabano M. Left Atrial Appendage Occlusion Without Fluoroscopy: Optimization by 4D Intracardiac Echocardiography. JACC Cardiovasc Interv. 2022 Aug 8;15(15):1592-1594. doi: 10.1016/j.jcin.2022.05.008. No abstract available. PMID 35926926
- [Background] Kim SS, Hijazi ZM, Lang RM, Knight BP. The use of intracardiac echocardiography and other intracardiac imaging tools to guide noncoronary cardiac interventions. J Am Coll Cardiol. 2009 Jun 9;53(23):2117-28. doi: 10.1016/j.jacc.2009.01.071. PMID 19497437
- [Background] Bartel T, Muller S, Biviano A, Hahn RT. Why is intracardiac echocardiography helpful? Benefits, costs, and how to learn. Eur Heart J. 2014 Jan;35(2):69-76. doi: 10.1093/eurheartj/eht411. Epub 2013 Oct 21. PMID 24144789
- [Background] Gianni C, Sanchez JE, Della Rocca DG, Al-Ahmad A, Horton RP, Di Biase L, Natale A. Intracardiac Echocardiography to Guide Catheter Ablation of Atrial Fibrillation. Card Electrophysiol Clin. 2021 Jun;13(2):303-311. doi: 10.1016/j.ccep.2021.03.009. Epub 2021 Apr 23. PMID 33990269
- [Background] D. Fornell, "First-in-Human Experience With Novel 4D ICE Catheter For Catheter Ablation and LAA Closure Procedures," 05 Aug 2021. [Online]. Available: https://www.dicardiology.com/content/first-human-experience-novel-4d-ice-catheter-catheter-ablation-and-laa-closure-procedures. [Accessed 18 Oct 2022].
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Bick RL, Frenkel EP. Clinical aspects of heparin-induced thrombocytopenia and thrombosis and other side effects of heparin therapy. Clin Appl Thromb Hemost. 1999 Oct;5 Suppl 1:S7-15. doi: 10.1177/10760296990050s103. PMID 10726030
- [Background] Cox B, Durieux ME, Marcus MA. Toxicity of local anaesthetics. Best Pract Res Clin Anaesthesiol. 2003 Mar;17(1):111-36. doi: 10.1053/bean.2003.0275. PMID 12751552
- [Background] Gruchalla RS. 10. Drug allergy. J Allergy Clin Immunol. 2003 Feb;111(2 Suppl):S548-59. doi: 10.1067/mai.2003.93. PMID 12592301
- [Background] Mertes PM, Laxenaire MC. Allergic reactions occurring during anaesthesia. Eur J Anaesthesiol. 2002 Apr;19(4):240-62. doi: 10.1017/s0265021502000418. PMID 12074414
- [Background] Morcos SK, Thomsen HS, Webb JA; Contrast Media Safety Committee of the European Society of Urogenital Radiology. Prevention of generalized reactions to contrast media: a consensus report and guidelines. Eur Radiol. 2001;11(9):1720-8. doi: 10.1007/s003300000778. PMID 11511894
- [Background] A. C. Lin and D. J. Wilber, Complications Associated With Radiofrequency Catheter Ablation, in Radiofrequency catheter ablation of cardiac arrhythmias: basic concepts and clinical applications, S. H. a. D. Wilber, Ed., Armonk, N.Y.: Futura Publishing Co. Inc., 2000, pp. 737-746
- [Background] Scheinman MM, Huang S. The 1998 NASPE prospective catheter ablation registry. Pacing Clin Electrophysiol. 2000 Jun;23(6):1020-8. doi: 10.1111/j.1540-8159.2000.tb00891.x. PMID 10879389
- [Background] Mar PL, Chong L, Perez A, Lakkireddy D, Gopinathannair R. Entrapment of diagnostic catheter within Advisor HD grid mapping catheter. J Cardiovasc Electrophysiol. 2021 Mar;32(3):860-861. doi: 10.1111/jce.14893. Epub 2021 Jan 28. PMID 33476457
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] Gerstenfeld EP, Guerra P, Sparks PB, Hattori K, Lesh MD. Clinical outcome after radiofrequency catheter ablation of focal atrial fibrillation triggers. J Cardiovasc Electrophysiol. 2001 Aug;12(8):900-8. doi: 10.1046/j.1540-8167.2001.00900.x. PMID 11513440
- [Background] Kovoor P, Ricciardello M, Collins L, Uther JB, Ross DL. Risk to patients from radiation associated with radiofrequency ablation for supraventricular tachycardia. Circulation. 1998 Oct 13;98(15):1534-40. doi: 10.1161/01.cir.98.15.1534. PMID 9769307
- [Background] Nahass GT. Fluoroscopy and the skin: implications for radiofrequency catheter ablation. Am J Cardiol. 1995 Jul 15;76(3):174-6. doi: 10.1016/s0002-9149(99)80053-8. No abstract available. PMID 7611155
- [Background] Calkins H, Niklason L, Sousa J, el-Atassi R, Langberg J, Morady F. Radiation exposure during radiofrequency catheter ablation of accessory atrioventricular connections. Circulation. 1991 Dec;84(6):2376-82. doi: 10.1161/01.cir.84.6.2376. PMID 1959193

RESULTS

PARTICIPANT FLOW:
Groups:
- NUVISION NAV Ultrasound Catheter: Participants with atrial arrhythmia and ventricular arrhythmia were enrolled and treated per investigator's standard of care while using the NUVISION NAV ultrasound catheter for ultrasound imaging and were followed-up until 7 days post-procedure. Atrial arrhythmia included subgroups as (a) scar-related atrial tachycardia (AT, including atypical atrial flutter)/ redo procedures resulting from previous atrial fibrillation ablation, (b) persistent atrial fibrillation (PsAF), and (c) paroxysmal atrial fibrillation (PVF). Ventricular arrhythmia included subgroups as (a) ventricular tachycardia (VT) including ischemic and non-ischemic VT and cardiomyopathy and idiopathic VT, and (b) premature ventricular complex (PVC).
Period: Overall Study
Arm/Group | NUVISION NAV Ultrasound Catheter
Started | 30
Participants Enrolled With Atrial Arrhythmia | 24
Participants Enrolled With Ventricular Arrhythmia | 6
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Completion of Imaging With the NUVISION NAV Ultrasound Catheter Without Resort to Non-study Mapping Catheter
Description: Percentage of participants with completion of imaging with the NUVISION NAV ultrasound catheter without resort to non-study mapping catheter were reported.
Time Frame: At Day 1
Population: Per Protocol (PP) analysis set included all enrolled participants who met the study eligibility criteria and in whom assessments were performed with the NUVISION NAV ultrasound catheter.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
Percentage of participants | 100.0 [88.4 to 100.0]

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Within 7 Days of Index Procedure Related to the NUVISION NAV Ultrasound Catheter
Description: Number of participants with SAEs within 7 days of index procedure related to the NUVISION NAV ultrasound catheter were reported. An AE was any untoward medical experience (sign, symptom, illness, abnormal laboratory value, or other medical event) occurring to a participant during the course of the study whether or not related to the investigational device. SAE was any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, was life-threatening experience, a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From day of index procedure (Day 1) up to 7 days
Population: Safety analysis set consisted of all enrolled participants who had undergone insertion of the NUVISION NAV ultrasound catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
Participants | 0

3. Secondary Outcome: Physician Assessment of Deployment, Maneuverability and Navigational Features With the NUVISION NAV Ultrasound Catheter During the Study Procedures
Description: Physician assessment of deployment, maneuverability and navigational features with the NUVISION NAV ultrasound catheter during the study procedures were reported. The physician's feedback was collected after each study procedure for each investigational catheter through a questionnaire-based survey consisting of 15 question/sub-question. Each survey question/sub-question included a response option with a Likert scale of 1 to 7 (1=poor and 7=excellent). A score of 4 on the Likert scales indicated the catheter met expectations or was comparable to other devices. Scores of greater than or equal to (>=) 4 were considered satisfaction.
Time Frame: Day 1
Population: PP analysis set included all enrolled participants who met study eligibility criteria and in whom assessments were performed with the NUVISION NAV ultrasound catheter. Here, 'n' (number analyzed) refers to number of participants analyzed for specified categories.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
Score on a scale
  Initial catheter introduction insert catheter into sheath | 7.0 [6.0 to 7.0]
  Advance catheter into heart | 7.0 [6.0 to 7.0]
  Visualize catheter on fluoroscopy | 7.0 [6.0 to 7.0]
  Catheter performance assessment deflection control | 7.0 [6.0 to 7.0]
  Deflection reach | 6.5 [5.0 to 7.0]
  Deflection degree (bi-directional) | 7.0 [5.0 to 7.0]
  Torqability | 7.0 [6.0 to 7.0]
  Ability to maintain torque | 7.0 [6.0 to 7.0]
  Tip rotation knob functionality | 7.0 [6.0 to 7.0]
  Catheter tip rotation | 7.0 [6.0 to 7.0]
  Ability to steer catheter within anatomy Manipulate catheter in right atrium (RA) | 7.0 [6.0 to 7.0]
  Manipulate catheter in left atrium (LA): number analyzed (Participants) | 12
  Manipulate catheter in left atrium (LA) | 7.0 [5.0 to 7.0]
  Ability to cross with catheter to LA: number analyzed (Participants) | 12
  Ability to cross with catheter to LA | 7.0 [6.0 to 7.0]
  Manipulate catheter in right ventricle (RV) | 7.0 [4.0 to 7.0]
  Manipulate catheter in left ventricle (LV): number analyzed (Participants) | 7
  Manipulate catheter in left ventricle (LV) | 7.0 [6.0 to 7.0]

4. Secondary Outcome: Physician Assessment of Imaging Quality Acquired With the NUVISION NAV Ultrasound Catheter During the Study Procedures
Description: Physician assessment of imaging quality acquired with the NUVISION NAV ultrasound catheter during the study procedures was reported. The quality of image acquired with NUVISION NAV ultrasound catheter and displayed by CARTO software was assessed through physician's feedback on 11 question/sub-questions. Each survey question/sub-question included a response option with a Likert scale of 1 to 7 (1=poor and 7=excellent). A score of 4 on the Likert scales indicated the catheter met expectations or was comparable to other devices. Scores of >=4 were considered satisfaction.
Time Frame: Day 1
Population: PP analysis set: all enrolled participants who met study eligibility criteria and in whom assessments were performed with NUVISION NAV ultrasound catheter. Here, 'N' (overall number of participants analyzed) refers to number of participants evaluable for this outcome measure; 'n' (number analyzed) refers to number of participants analyzed for specified categories.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 29
Score on a scale
  Contouring, value of drawing CARTOSOUND contours on 2D ultrasound image: number analyzed (Participants) | 26
  Contouring, value of drawing CARTOSOUND contours on 2D ultrasound image | 7.0 [5.0 to 7.0]
  On dual-plane: number analyzed (Participants) | 26
  On dual-plane | 6.0 [5.0 to 7.0]
  On multi-plane: number analyzed (Participants) | 26
  On multi-plane | 6.0 [5.0 to 7.0]
  General did CARTO integration help you to orient in multi-plane?: number analyzed (Participants) | 28
  General did CARTO integration help you to orient in multi-plane? | 6.0 [4.0 to 7.0]
  Did CARTO integration help you to orient in 4D?: number analyzed (Participants) | 28
  Did CARTO integration help you to orient in 4D? | 6.0 [4.0 to 7.0]
  Did image on CARTO screen change as predicted when deflecting in anterior and posterior directions?: number analyzed (Participants) | 25
  Did image on CARTO screen change as predicted when deflecting in anterior and posterior directions? | 6.0 [5.0 to 7.0]
  How useful was the 'store clip' on CARTO?: number analyzed (Participants) | 24
  How useful was the 'store clip' on CARTO? | 6.0 [4.0 to 7.0]
  Was troubleshooting information provided by the system helpful?: number analyzed (Participants) | 15
  Was troubleshooting information provided by the system helpful? | 6.0 [5.0 to 7.0]
  Was the green tip overlay on the different planes useful? | 6.0 [6.0 to 7.0]
  Was the indication of Live vs. Review Modes clear enough? | 6.0 [6.0 to 7.0]
  How useful was intracardiac echocardiography (ICE) guidance for performing the transseptal puncture?: number analyzed (Participants) | 26
  How useful was intracardiac echocardiography (ICE) guidance for performing the transseptal puncture? | 7.0 [6.0 to 7.0]

5. Secondary Outcome: Physicians Overall Feedback on the NUVISION NAV Ultrasound Catheter During the Study Procedures
Description: Physicians overall feedback on the NUVISION NAV ultrasound catheter during the study procedure was reported. The overall feedback on the NUVISION NAV ultrasound catheter was assessed through physician's feedback on 3 question/sub-questions. Each survey question/sub-question included a response option with a Likert scale of 1 to 7 (1=poor and 7=excellent). A score of 4 on the Likert scales indicated the catheter met expectations or was comparable to other devices. Scores of >=4 were considered satisfaction. TEE is transesophageal echocardiography.
Time Frame: Day 1
Population: PP analysis set: all enrolled participants who met study eligibility criteria and in whom assessments were performed with NUVISION NAV ultrasound catheter. Here, 'n' (number analyzed) refers to number of participants analyzed for specified categories.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
Score on a scale
  Do you think that the NUVISION NAV ultrasound catheter is an acceptable alternative to TEE?: number analyzed (Participants) | 29
  Do you think that the NUVISION NAV ultrasound catheter is an acceptable alternative to TEE? | 7.0 [6.0 to 7.0]
  What is your overall satisfaction of the NUVISION NAV ultrasound catheter? | 7.0 [6.0 to 7.0]
  Would you recommend the NUVISION NAV ultrasound catheter to fellow physicians? | 7.0 [4.0 to 7.0]

6. Secondary Outcome: Number of Serious Adverse Events (SAEs) Excluding NUVISION NAV Ultrasound Catheter Related SAE Within 7 Days of Index Procedure
Description: Number of SAEs excluding NUVISION NAV ultrasound catheter related SAE within 7 days of index procedure was reported. AE was any untoward medical experience (sign, symptom, illness, abnormal laboratory value, or other medical event) occurring to a participant during the course of the study whether or not related to the investigational device. SAE was any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, was life-threatening experience, a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From day of index procedure (Day 1) up to 7 days
Population: as for outcome 2
Measure: Number; unit: SAEs
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
SAEs | 2 [0.8 to 22.1]

7. Secondary Outcome: Number of Participants With Non-serious Adverse Events Within 7 Days of Index Procedure Related to the NUVISION NAV Ultrasound Catheter
Description: Number of participants with non-serious adverse events within 7 days of index procedure related to the NUVISION NAV ultrasound catheter were reported. AE was any untoward medical experience (sign, symptom, illness, abnormal laboratory value, or other medical event) occurring to a participant during the course of the study whether or not related to the investigational device.
Time Frame: From day of index procedure (Day 1) up to 7 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NUVISION NAV Ultrasound Catheter
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 7 days after index procedure on Day 1
Description: Safety analysis set consisted of all enrolled participants who had undergone insertion of the NUVISION NAV ultrasound catheter.
Arm/Group | NUVISION NAV Ultrasound Catheter
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NUVISION NAV Ultrasound Catheter (N=30)
Complete Atrioventricular block (Cardiac disorders) | 1
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NUVISION NAV Ultrasound Catheter (N=30)
Pericardial Effusion (Cardiac disorders) | 1
Delayed Wound Healing (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications and/or presentation of clinical investigation results will be coordinated and governed between Biosense Webster, Inc., the clinical investigation author(s) and if applicable local law. Authorship will be determined prior to development of any manuscript.

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT05970120/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT05970120/SAP_001.pdf